CLINICAL TRIAL: NCT02542696
Title: An Open-Label, Phase 3 Study Examining the Long-Term Safety, Tolerability and Efficacy of APL-130277 in Levodopa Responsive Patients With Parkinson's Disease Complicated by Motor Fluctuations ("OFF" Episodes)
Brief Title: Open-Label Phase 3 Study to Examine the Long-Term Safety, Tolerability and Efficacy of APL-130277 for the Acute Treatment of "OFF" Episodes in Patients With Parkinson's Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CTH-301; 2016-000637-43 (EudraCT Number)
Record Dates: First submitted 2015-09-03; First posted 2015-09-07 (Estimated); Results first posted 2023-11-22 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-10

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Apomorphine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- APL-130277 (Experimental): APL-130277 sublingual thin film (10 mg, 15 mg, 20 mg, 25 mg, 30 mg and 35 mg)
  Interventions: Drug: APL-130277

INTERVENTIONS:
Drug: APL-130277 — Used to treat up to 5 "OFF" episodes per day
  Other Names: Apomorphine Hydrochloride, Sublingual Thin Film

SUMMARY:
An Open-Label Phase 3 Study to Examine the Long-Term Safety, Tolerability and Efficacy of APL-130277 for the Acute Treatment of "OFF" Episodes in Patients With Parkinson's Disease

ELIGIBILITY:
De Novo Subjects Inclusion Criteria

1. Male or female ≥ 18 years of age.
2. Clinical diagnosis of Idiopathic PD, consistent with UK Brain Bank Criteria (excluding the "more than one affected relative" criterion)
3. Clinically meaningful response to L-Dopa as determined by the Investigator.
4. Receiving stable doses of L-Dopa/carbidopa (immediate or CR) administered at least 4 times per day OR Rytary™ administered at least 3 times per day, for at least 4 weeks before the initial Screening Visit (SV1). Adjunctive PD medication regimens must be maintained at a stable dose for at least 4 weeks prior to the initial Screening Visit (SV1) with the exception that MAO-B inhibitors must be maintained at a stable level for at least 8 weeks prior to the initial Screening Visit (SV1).
5. No planned medication change(s) or surgical intervention anticipated during the course of study.
6. Subject must experience at least one well defined "OFF" episode per day with a total daily "OFF" time duration of ≥ 2 hours during the waking day, based on patient self-assessment.
7. Subject and/or caregiver must be trained in performing home dosing diary assessments of the motor state and must be able to recognize "ON" and "OFF" states.
8. Stage III or less on the modified Hoehn and Yahr scale in the "ON" state.
9. MMSE score > 25.
10. If female and of childbearing potential, must agree to be sexually abstinent or use one of the following highly effective methods of birth control:

    * Hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants);
    * Intrauterine contraceptive system;
    * Surgical sterilization or partner sterile (must have documented proof); AND

    One of the following effective methods of birth control:
    * Male/female condom;
    * Cervical cap with spermicide;
    * Diaphragm with spermicide;
    * Contraceptive sponge.
11. Male subjects must be either surgically sterile, agree to be sexually inactive or use a double-barrier method of birth control (eg, condom and diaphragm with spermicide, condom with cervical cap and spermicide) from first study drug administration until 90 days after final drug administration.
12. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures.
13. Able to understand the consent form, and to provide written informed consent.

De Novo Subjects Exclusion Criteria -

1. Atypical or secondary parkinsonism.
2. Previous treatment with any of the following: a neurosurgical procedure for PD; continuous s.c. apomorphine infusion; Duodopa/Duopa; or APL-130277.
3. Treatment with any form of s.c. apomorphine within 7 days prior to the second Screening Visit (SV2). Patients that stopped s.c. apomorphine for any reason other than systemic safety concerns or lack of efficacy may be considered.
4. Contraindications to APOKYN®, or hypersensitivity to apomorphine hydrochloride or any of the ingredients of APOKYN® (notably sodium metabisulfite).
5. Female who is pregnant or lactating.
6. Participation in a clinical trial within 30 days prior to the initial Screening Visit (SV1).
7. Receipt of any investigational (ie, unapproved) medication within 30 days prior to the initial Screening Visit (SV1).
8. Currently taking selective 5HT3 antagonists (ie, ondansetron, granisetron, dolasetron, palonosetron, alosetron), dopamine antagonists (excluding quetiapine or clozapine) or dopamine depleting agents.
9. Drug or alcohol dependency in the past 12 months.
10. Subject has a history of malignancy within 5 years prior to the Screening visit, except for adequately treated basal cell or squamous cell skin cancer or in situ cervical cancer. Pituitary tumors of any duration are excluded.
11. Clinically significant medical, surgical, or laboratory abnormality in the opinion of the Investigator.
12. Major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis, or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
13. History of clinically significant hallucinations during the past 6 months.
14. History of clinically significant impulse control disorder(s).
15. Dementia that precludes providing informed consent or would interfere with participation in the study.
16. Current suicidal ideation within one year prior to the second Screening Visit (SV2) as evidenced by answering "yes" to Questions 4 or 5 on the suicidal ideation portion of the C-SSRS or attempted suicide within the last 5 years.
17. Donation of blood or plasma in the 30 days prior to first dosing.
18. Presence of canker or mouth sores in the 30 days prior to the initial Screening Visit (SV1), or other clinically significant oral pathology in the opinion of the Investigator. The Investigator should follow-up with an appropriate specialist on any finding, if indicated, before enrolling a patient into the study.

Rollover Subjects Inclusion Criteria

1. Completion of any of the following studies: CTH-201, CTH-203, CTH-300, or CTH 302; and, in the opinion of the Investigator, would benefit from continued treatment with APL 130277.
2. No major changes in concomitant PD medications since completion of any of the following studies: CTH-201, CTH-203, CTH-300, or CTH 302. Any change in PD medications since the previous study should be discussed with the Medical Monitor to determine subject eligibility in the current study.
3. If female and of childbearing potential, must agree to be sexually abstinent or use one of the following highly effective methods of birth control:

   * Hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants);
   * Intrauterine contraceptive system;
   * Surgical sterilization or partner sterile (must have documented proof); AND

   One of the following effective methods of birth control:
   * Male/female condom;
   * Cervical cap with spermicide;
   * Diaphragm with spermicide;
   * Contraceptive sponge.
4. Male subjects must be either surgically sterile, agree to be sexually inactive or use a double-barrier method of birth control (eg, condom and diaphragm with spermicide, condom with cervical cap and spermicide) from first study drug administration until 90 days after final drug administration.
5. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures.
6. Able to understand the consent form, and to provide written informed consent.

Rollover Subjects Exclusion Criteria

1. Female who is pregnant or lactating.
2. Presence of any major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis (including clinically significant hallucinations during the past 6 months) or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation unsafe or make treatment compliance difficult.
3. Presence of any clinically significant medical (including but not limited to CNS, cardiovascular, hepatic, pulmonary, metabolic, or renal events), surgical, or laboratory abnormality that would make study participation unsafe or make treatment compliance difficult. Clinical significance to be determined by the Investigator.
4. Receipt of any investigational (ie, unapproved) medication or participation in any clinical trial of an investigational product since completing a previous study using APL 130277.
5. Development of canker or mouth sores within 14 days of completing a previous study using APL-130277. For other clinically significant oral pathology, the Investigator should follow-up with an appropriate specialist on any finding, if indicated, before enrolling such a subject into the study. Clinical significance to be determined by the Investigator. The eligibility of subjects who have experienced AEs related to the oral cavity during the previous study using APL-130277, should be reviewed with the medical monitor and approval obtained.
6. Current suicidal ideation within one year of the screening visit, as evidenced by answering "yes" to Question 4 or 5 on the suicidal ideation portion of the C SSRS at Screening or attempted suicide within 5 years.

CTH-301 Completer Subjects Inclusion Criteria

1. Completion of the CTH-301 study under protocol version 3.00, and in the opinion of the Investigator, would benefit from continued treatment with APL 130277.
2. If female and of childbearing potential, must agree to be sexually abstinent or use one of the following highly effective methods of birth control:

   * Hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants);
   * Intrauterine contraceptive system;
   * Surgical sterilization or partner sterile (must have documented proof); AND

   One of the following effective methods of birth control:
   * Male/female condom;
   * Cervical cap with spermicide;
   * Diaphragm with spermicide;
   * Contraceptive sponge.
3. Male subjects must be either surgically sterile, agree to be sexually inactive or use a double-barrier method of birth control (eg, condom and diaphragm with spermicide, condom with cervical cap and spermicide) from first study drug administration until 90 days after final drug administration.
4. Willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study-related procedures.
5. Able to understand the consent form, and to provide written informed consent.

CTH-301 Completer Subjects Exclusion Criteria

1. Female who is pregnant or lactating.
2. Presence of any major psychiatric disorder including, but not limited to, dementia, bipolar disorder, psychosis (including clinically significant hallucinations during the past 6 months) or any disorder that, in the opinion of the Investigator, requires ongoing treatment that would make study participation in unsafe or make treatment compliance difficult.
3. Presence of any clinically significant medical (including but not limited to CNS, cardiovascular, hepatic, pulmonary, metabolic, or renal events), surgical, or laboratory abnormality that would make study participation unsafe or make treatment compliance difficult. Clinical significance to be determined by the Investigator.
4. Receipt of any investigational (ie, unapproved) medication or participation in any clinical trial since completing the CTH 301 study.
5. Development of canker or mouth sores since completing the CTH 301 study. For other clinically significant oral pathology, the Investigator should follow-up with an appropriate specialist on any finding, if indicated, before enrolling such a patient into the study. Clinical significance to be determined by the Investigator.
6. Current suicidal ideation as evidenced by answering "yes" to Question 4 or 5 on the suicidal ideation portion of the C-SSRS at the Screening Visit Phase 2 (SVP2).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 496 (Actual)
Dates: Start 2015-08-31 (Actual); Primary Completion 2022-11-08 (Actual); Study Completion 2022-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: CNS Medical Director, Study Director — Sumitomo Pharma America, Inc.
Locations (70):
- United States (48):
  - University of Alabama Birmingham, Birmingham, Alabama
  - Muhammed Ali Parkinson and Movement Disorder Center/Barrow Neurological Institute, Phoenix, Arizona
  - Movement Disorders Center of Arizona, Scottsdale, Arizona
  - Clinical Trials, Inc., Little Rock, Arkansas
  - The Parkinson's and Movement Disorder Institute, Fountain Valley, California
  - UC Irvine Health Gottschalk Medical Plaza, Irvine, California
  - Keck Medical Center at USC, Los Angeles, California
  - University of Colorado School of Medicine, Aurora, Colorado
  - MedStar Georgetown University Hospital, Washington D.C., District of Columbia
  - Parkinsons Disease and Movement Disorders Center, Boca Raton, Florida
  - University of Miami, Miller School of Medicine, Miami, Florida
  - Parkinson's Disease Treatment Center of Southwest Florida, Port Charlotte, Florida
  - Suncoast Neuroscience Associates Inc., St. Petersburg, Florida
  - USF Parkinson's Disease and Movement Disorder Center, Tampa, Florida
  - Emory University Department of Neurology, Atlanta, Georgia
  - GRU Movement Disorders, Augusta, Georgia
  - Northwestern University, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - NorthShore Neurological Institute B043D, Glenview, Illinois
  - Central DuPage Hospital - Neurodegenerative Clinic - Movement Disorders Center, Winfield, Illinois
  - University of Iowa Dept. of Neurology, Iowa City, Iowa
  - Kansas University Medical Center-Department of Neurology, Kansas City, Kansas
  - University of Kentucky, Lexington, Kentucky
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University, Baltimore, Maryland
  - Michigan State University - Dept. of Neurology, East Lansing, Michigan
  - QUEST Research Institute, Farmington Hills, Michigan
  - Henry Ford Hospital, West Bloomfield, Michigan
  - Park Nicolet Institute - Stuthers Parkinson's Center, Golden Valley, Minnesota
  - SUNY Downstate Medical Center, Department of Neurology, Brooklyn, New York
  - Bendheim Parkinson's and Movement Disorder Center (Mount Sinai Medical Center), New York, New York
  - Columbia University Medical Center - Neurological Institute, Movement Disorders, New York, New York
  - Duke University - Movement Disorders Clinic, Durham, North Carolina
  - Raleigh Neurology Associates, P.A., Raleigh, North Carolina
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University Wexner Medical Center, Columbus, Ohio
  - UT Gardner-McMaster Parkinson's Center, Toledo, Ohio
  - The Movement Disorder Clinic of Oklahoma, Tulsa, Oklahoma
  - Jefferson University Hospital Philadelphia, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - Houston Methodist Neurological Institute, Houston, Texas
  - East Texas Medical Center, Tyler, Texas
  - University of Virginia Adult Neurology, Charlottesville, Virginia
  - Sentara Neuroscience Institute, Virginia Beach, Virginia
  - Evergreen Health, Kirkland, Washington
  - Swedish Neuroscience Research, Seattle, Washington
- Austria (2):
  - Medical University Innsbruck Neurology Department, Innsbruck
  - Wilhelminenspital Department of Neurology, Vienna
- UHN Toronto Western Hospital, Toronto, Ontario, Canada
- Centre d'Investigation Clinique, CIC 1436, CHU Purpan, Toulouse, France
- Germany (2):
  - St. Josef-Hospital, Klinikum der Ruhr-Universitaet-Bochum, Neurologische Klinik, Bochum
  - Universitätsklinikum Ulm Neurologisches Studienzentrum im RKU, Ulm
- Italy (4):
  - Ospedali Riuniti di Ancona, Ancona
  - Centro Ricerche San Raffaele, Cassino
  - Aging Research Center, Ce.S.I. University Foundation, Chieti-Pescara Behavioural Neurology & Movement Disorders Unit, Chieti
  - IRCCS San Raffaele Pisana - Clinical Trial Center, Rome
- Spain (2):
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Universitari General de Catalunya, Sant Cugat Del Vallés
- United Kingdom (10):
  - Kings College, The Maurice Wohl Neuroscience Institute, London, Greater London
  - Manchester University, Salford, Greater Manchester
  - Newcastle University, Newcastle upon Tyne, Northumberland
  - Forth Valley Royal Hospital, Larbert, Stirlingshire
  - Fairfield General Hospital, Bury
  - Royal Devon & Exeter NHS Foundation Trust, Exeter
  - Queen Elizabeth University Hospital, Glasgow
  - Leeds Teaching Hospitals NHS Trust, Leeds
  - Imperial College Healthcare Trust NHS, London
  - Plymouth University, Plymouth

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | APL-130277
Started | 496
Titration Full Analysis Population | 449
LTS Phase Full Analysis Population | 426
Completed | 120
Not Completed | 376
Not completed — Adverse Event | 167
Not completed — Lack of Efficacy | 26
Not completed — Lost to Follow-up | 6
Not completed — Withdrawal by Subject | 104
Not completed — Protocol Violation | 5
Not completed — Death | 8
Not completed — DECREASED OFF TIME | 1
Not completed — DID NOT MEET CRITERIA FOR CONTINUATION | 1
Not completed — ELIGIBILITY CRITERIA NOT MET | 8
Not completed — MEDICAL HISTORY | 1
Not completed — PATIENT WITHDRAWN DURING TITRATION AS COULD NOT TITRATE DRUG TO GET RESPONSE OF "ON" FROM PATIENT | 1
Not completed — PROGRESSION OF PARKINSON'S DISEASE | 5
Not completed — SITE UNABLE TO COMPLY WITH PROTOCOL | 2
Not completed — SPONSOR DECISION | 3
Not completed — STUDY TERMINATED BY SPONSOR | 36
Not completed — SUBJECT DECISION | 2

BASELINE CHARACTERISTICS:
Arm/Group | APL-130277
Number analyzed (Participants) | 496
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 239
  >=65 years | 257
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.4 (8.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 163
  Male | 333
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39
  Not Hispanic or Latino | 457
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1
  Asian | 4
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 10
  White | 478
  More than one race | 0
  Unknown or Not Reported | 2
ON State Modified Hoehn and Yahr Score [Count of Participants; unit: Participants] — The scale has been used for the staging of the functional disability associated with Parkinson's disease. STAGE 0 = No signs of disease. STAGE 1 = Unilateral disease. STAGE 1.5 = Unilateral plus axial involvement. STAGE 2 = Bilateral disease, without impairment of balance. STAGE 2.5 = Mild bilateral disease, with recovery on pull test. STAGE 3 = Mild to moderate bilateral disease; some postural instability; physically independent. STAGE 4 = Severe disability; still able to walk or stand unassisted. STAGE 5 = Wheelchair bound or bedridden unless aided.
  Participants
    0 | 2
    1 | 12
    1.5 | 9
    2 | 243
    2.5 | 53
    3 | 42
    4 | 1
    Missing | 134
Age, Customized [Count of Participants; unit: Participants]
  <65 years | 239
  >=65 years and <75 years | 197
  >=75 years | 60
Baseline Height (cm) [Mean (Standard Deviation); unit: cm] — Population: some subjects had missing height measurement
  cm
    number analyzed (Participants) | 488
    (all) | 172.01 (9.754)
Baseline Weight (kg) [Mean (Standard Deviation); unit: kg] — Population: some subjects had missing weight at baseline
  kg
    number analyzed (Participants) | 492
    (all) | 82.14 (18.740)
Baseline BMI (kg/m^2) [Mean (Standard Deviation); unit: kg/m^2] — Population: some subjects had missing BMI value at baseline
  kg/m^2
    number analyzed (Participants) | 487
    (all) | 27.654 (5.5287)
Country [Count of Participants; unit: Participants]
  Aut | 4
  Can | 7
  Deu | 23
  Esp | 11
  Gbr | 41
  Ita | 19
  United States | 391
Baseline MDS-UPDRS Part III Score [Mean (Standard Deviation); unit: Score] — The summary score used here is Part III motor examination score. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4 (0=normal, 1=slight, 2=mild, 3= moderate, and 4=severe). The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome). Population: based on subjects with data only
  Score
    number analyzed (Participants) | 426
    (all) | 43.0 (14.85)
Screening MDS-UPDRS Part III Score [Mean (Standard Deviation); unit: Score] — The summary score used here is Part III motor examination score. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4 (0=normal, 1=slight, 2=mild, 3= moderate, and 4=severe). The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome). Population: Based on subjects with data only
  Score
    number analyzed (Participants) | 367
    (all) | 42.0 (14.55)
Mini-Mental State Examination Total Score [Count of Participants; unit: Participants] — Mini-Mental State Examination Total Score is a global assessment of cognitive status. Severe cognitive impairment: 0-17 Mild cognitive impairment: 18-23 No cognitive impairment: 24-30
  Participants
    <26 | 3
    26 | 30
    27 | 38
    28 | 53
    29 | 114
    30 | 183
    Missing | 75
Baseline MDS-UPDRS Part I Score [Mean (Standard Deviation); unit: Score] — MDS-UPDRS Part I Score measures nonmotor experiences of daily living: 13 items. Score range: 0-52, 10 and below is mild, 22 and above is severe. Population: Only subjects with data were summarized
  Score
    number analyzed (Participants) | 492
    (all) | 11.0 (5.42)
Baseline MDS-UPDRS Part II Score [Mean (Standard Deviation); unit: Score] — MDS-UPDRS Part II Score measures motor experiences of daily living: 13 items. Score range: 0-52, 12 and below is mild, 30 and above is severe. Population: based on subjects with data only
  Score
    number analyzed (Participants) | 492
    (all) | 14.6 (7.15)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety and Tolerability Data Collected, Based on Number of Participants With Adverse Events in the LTS Phase
Description: Number of Participants (%) with Adverse Events in the LTS Phase
Time Frame: up to approximately 3 years
Population: Based on Long Term Safety Full Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | APL-130277
Number analyzed (Participants) | 426
Participants | 365

2. Secondary Outcome: The Percentage of Instances Where a Full "ON" Response Was Achieved Within 30 Minutes After Self-administration of Study Medication at Week 24 Visit (LTS V4) of the LTS Phase Based on the Home Dosing Diary Entries.
Description: The percentage of instances where a full "ON" response was achieved
Time Frame: Week 24
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: percentage of instances
Arm/Group | APL-130277
Number analyzed (Participants) | 167
percentage of instances | 80.7 (32.55)

3. Secondary Outcome: The Percentage of Instances Where a Full "ON" Response Was Achieved Within 30 Minutes After Self-administration of Study Medication at Week 36 Visit (LTS V5) of the LTS Phase Based on the Home Dosing Diary Entries.
Time Frame: Week 36
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: percentage of instances
Arm/Group | APL-130277
Number analyzed (Participants) | 80
percentage of instances | 87.3 (28.70)

4. Secondary Outcome: The Percentage of Instances Where a Full "ON" Response Was Achieved Within 30 Minutes After Self-administration of Study Medication at Week 48 Visit (LTS V6) of the LTS Phase Based on the Home Dosing Diary Entries.
Time Frame: Week 48
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: percentage of instances
Arm/Group | APL-130277
Number analyzed (Participants) | 70
percentage of instances | 84.1 (30.74)

5. Secondary Outcome: Percentage of Subjects With a Subject-rated Full "ON" Response Within 30 Minutes at Week 24 Visit (LTS V4) of the LTS Phase.
Time Frame: Week 24
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Number; unit: percent of participants
Arm/Group | APL-130277
Number analyzed (Participants) | 224
percent of participants | 77.2

6. Secondary Outcome: Percentage of Subjects With a Subject-rated Full "ON" Response Within 30 Minutes at Week 36 Visit (LTS V5) of the LTS Phase.
Time Frame: Week 36
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Number; unit: percent of participants
Arm/Group | APL-130277
Number analyzed (Participants) | 112
percent of participants | 83.9

7. Secondary Outcome: Percentage of Subjects With a Subject-rated Full "ON" Response Within 30 Minutes at Week 48 Visit (LTS V6) of the LTS Phase.
Time Frame: Week 48
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Number; unit: percent of participants
Arm/Group | APL-130277
Number analyzed (Participants) | 90
percent of participants | 84.4

8. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 15 Minutes After Dosing at Week 24 Visit (LTS V4) of the LTS Phase.
Description: The summary score used here is Part III motor examination score. Higher MDS-UPDRS scores reflect worse motor function. MDS-UPDRS III is a total of 18 questions with 33 individual items, each item ranges from 0-4 (0=normal, 1=slight, 2=mild, 3= moderate, and 4=severe). The MDS-UPDRS III motor score is the summation of all these 33 individual item scores, and hence ranges from 0-132. Score drops over time imply improvement in motor function (higher values represent a worse outcome).
Time Frame: Week 24, 15 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- APL-103277: APL-130277 sublingual thin film (10 mg, 15 mg, 20 mg, 25 mg, 30 mg and 35 mg)
Arm/Group | APL-103277
Number analyzed (Participants) | 223
Units on a scale | -14.2 (11.91)

9. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 30 Minutes After Dosing at Week 24 Visit (LTS V4) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 24, 30 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 222
Units on a scale | -22.1 (13.04)

10. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 60 Minutes After Dosing at Week 24 Visit (LTS V4) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 24, 60 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 221
Units on a scale | -21.0 (13.34)

11. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 90 Minutes After Dosing at Week 24 Visit (LTS V4) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 24, 90 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 48
Units on a scale | -16.9 (13.58)

12. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 15 Minutes After Dosing at Week 36 Visit (LTS V5) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 36, 15 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 111
Units on a scale | -11.7 (10.48)

13. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 30 Minutes After Dosing at Week 36 Visit (LTS V5) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 36, 30 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 110
Units on a scale | -22.3 (12.22)

14. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 60 Minutes After Dosing at Week 36 Visit (LTS V5) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 36, 60 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 112
Units on a scale | -21.3 (13.54)

15. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 90 Minutes After Dosing at Week 36 Visit (LTS V5) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 36, 90 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 54
Units on a scale | -13.3 (13.11)

16. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 15 Minutes After Dosing at Week 48 Visit (LTS V6) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 48, 15 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 90
Units on a scale | -13.3 (10.17)

17. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 30 Minutes After Dosing at Week 48 Visit (LTS V6) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 48, 30 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 90
Units on a scale | -23.2 (12.44)

18. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 60 Minutes After Dosing at Week 48 Visit (LTS V6) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 48, 60 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 90
Units on a scale | -22.3 (13.35)

19. Secondary Outcome: Mean Change From Pre-dose in MDS-UPDRS Part III Motor Examination (MDS UPDRS MOTOR) Score at 90 Minutes After Dosing at Week 48 Visit (LTS V6) of the LTS Phase.
Description: as for outcome 8
Time Frame: Week 48, 90 mins after dosing
Population: Based on the number of subjects who provided data at the specified timepoint in the analysis population
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | APL-103277
Number analyzed (Participants) | 48
Units on a scale | -16.6 (10.93)

ADVERSE EVENTS:
Time Frame: Up to approximately 3 years for Long Term Safety Phase, including up to approximately 22 weeks for titration phase.
Arm/Group | APL-130277
All-Cause Mortality (participants affected / at risk) | 8/496
Serious Adverse Events (participants affected / at risk) | 64/496
Other Adverse Events (participants affected / at risk) | 319/496
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (N=496)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 3 (3)
Angina unstable (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Atrioventricular block complete (Cardiac disorders) | 1 (1)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Bradyarrhythmia (Cardiac disorders) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 3 (3)
Cardio-respiratory arrest (Cardiac disorders) | 1 (1)
Coronary artery stenosis (Cardiac disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Sinus node dysfunction (Cardiac disorders) | 1 (1)
Retinal artery occlusion (Eye disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Duodenitis (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1)
Lip blister (Gastrointestinal disorders) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 2 (2)
Chest pain (General disorders) | 1 (2)
Drowning (General disorders) | 2 (2)
General physical health deterioration (General disorders) | 1 (1)
Hepatitis toxic (Hepatobiliary disorders) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (3)
Corona virus infection (Infections and infestations) | 2 (2)
Kidney infection (Infections and infestations) | 1 (1)
Oral candidiasis (Infections and infestations) | 1 (1)
Osteomyelitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 5 (5)
Psoas abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Septic shock (Infections and infestations) | 1 (1)
Streptococcal sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 4 (6)
Urosepsis (Infections and infestations) | 1 (1)
Wound infection (Infections and infestations) | 1 (1)
Adjacent segment degeneration (Injury, poisoning and procedural complications) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 5 (5)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1)
Fractured sacrum (Injury, poisoning and procedural complications) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Rib fracture (Injury, poisoning and procedural complications) | 2 (2)
Spinal compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon injury (Injury, poisoning and procedural complications) | 1 (1)
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1)
Carbon dioxide increased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Arthropathy (Musculoskeletal and connective tissue disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (2)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Bone cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Prostate cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Autonomic nervous system imbalance (Nervous system disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Coma (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Myelopathy (Nervous system disorders) | 1 (1)
Neuropathy peripheral (Nervous system disorders) | 1 (1)
Parkinson's disease (Nervous system disorders) | 2 (2)
Subarachnoid haematoma (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Adjustment disorder with mixed anxiety and depressed mood (Psychiatric disorders) | 1 (2)
Depression (Psychiatric disorders) | 1 (1)
Dopamine dysregulation syndrome (Psychiatric disorders) | 1 (1)
Mental status changes (Psychiatric disorders) | 1 (1)
Psychotic disorder (Psychiatric disorders) | 1 (1)
Substance-induced psychotic disorder (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder neck obstruction (Renal and urinary disorders) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 1 (1)
Cystitis haemorrhagic (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
Obstructive uropathy (Renal and urinary disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural thickening (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | APL-130277 (N=496)
Lip swelling (Gastrointestinal disorders) | 27 (36)
Mouth ulceration (Gastrointestinal disorders) | 28 (37)
Nausea (Gastrointestinal disorders) | 136 (197)
Oral mucosal erythema (Gastrointestinal disorders) | 43 (60)
Stomatitis (Gastrointestinal disorders) | 25 (39)
Fatigue (General disorders) | 35 (48)
Fall (Injury, poisoning and procedural complications) | 44 (63)
Dizziness (Nervous system disorders) | 52 (70)
Dyskinesia (Nervous system disorders) | 34 (47)
Headache (Nervous system disorders) | 31 (43)
Somnolence (Nervous system disorders) | 57 (81)
Yawning (Respiratory, thoracic and mediastinal disorders) | 55 (99)
Vomiting (Gastrointestinal disorders) | 25 (33)
Orthostatic hypotension (Vascular disorders) | 26 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In the event the Study is part of a multi-center study, the first publication of the results of the Study shall be made in conjunction with the results of other participating study sites as a multi-center publication; provided however, if a multi-center publication is not forthcoming within twenty-four (24) months following completion of the Study at all sites, Institution and Investigator shall be free to publish.

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/96/NCT02542696/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-29): https://cdn.clinicaltrials.gov/large-docs/96/NCT02542696/SAP_001.pdf